CLINICAL TRIAL: NCT02555956
Title: Subthreshold Double Frequency Nd. YAG Grid Laser for Diffuse Diabetic Maculopathy
Brief Title: Grid Laser for Diffuse Diabetic Maculopathy
Acronym: MMG
Status: Completed | Type: Observational
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Jamshed Ahmed, Assistant Professor, Dow University of Health Sciences
Other Study IDs: Macular Grid Laser
Record Dates: First submitted 2015-08-06; First posted 2015-09-22 (Estimated); Last update posted 2015-09-22 (Estimated); Status verified 2015-09

CONDITIONS: Diabetic Macular Edema
Keywords: Macular grid; Subthreshold; diabetic macular edema; decrease in visual acuity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Diabetic related complications are increasing day by day due to increse in the number of diabetic patients all over the world. Diabetic macular edema is one of them and a major cause of vision imparment. Various kind of treatment modalities are preent to treat this coplication. Grid laser is one treatment modality. Laser phtocoagulation is a destrictive procedure.Laser power if kept to aminimum can get the desired results without severe destruction to the retina . In this study, the investigators are going to document the effect of minimal grid laser tn loss o overcome the visioe to diabetic macular edema.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic patients with macular edema.
* both sexes
* conset to participate.

Exclusion Criteria:

* focal edema.
* patients requiring only the focal laser.
* patients with proferative diabetic retinopathy.
* Patients with ischaemic maculopathy on fundus fluorescein angiography.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetic patients having diffuse diabetic macular edema.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2012-04; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Improvement of visual acuity after grid laser | 6 week
  Visual acuity will be mesured pre laser and 06 weeks post laser

SECONDARY OUTCOMES:
Complication | during first six weeks after laser
  Patiens willbe asked and examined for any potentiail anticipated complication.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Jamshed Ahmed, FCPS, Principal Investigator — Dow university of health sciences, karachi; Jamshed Ahmed, FCPS, Principal Investigator — Dow University of Health Sciences
Locations (1):
- Dow universty Hospital,Dow international Medical college, Karachi, Sindh, Pakistan